CLINICAL TRIAL: NCT02601222
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Trials to Evaluate the Efficacy and Safety of Runzao Zhiyang Capsule in Treating Chronic Eczema
Brief Title: Efficacy and Safety of Runzao Zhiyang Capsule to Treat Chronic Eczema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Tongjitang Pharmaceutical Co.,Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z-RZZY-JN-RS
Record Dates: First submitted 2015-10-09; First posted 2015-11-10 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Eczema
Keywords: chronic eczema; efficacy and safety; Runzao zhiyang capsule

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Runzao zhiyang capsule (Experimental): Runzao zhiyang capsule: 4 pills each time, 3 times a day, oral， Urea Cream (topical application, apply to the affected area and gently rub) 2 times a day.
  Interventions: Drug: Runzao zhiyang capsule; Drug: Urea cream
- Runzaozhiyang capsule agent simulation (Placebo Comparator): Runzaozhiyang capsule agent simulation:4 pills each time, 3 times a day, oral, Urea Cream (topical application, apply to the affected area and gently rub) 2 times a day.
  Interventions: Drug: Runzaozhiyang capsule agent simulation; Drug: Urea cream

INTERVENTIONS:
Drug: Runzao zhiyang capsule — Runzao zhiyang capsule：4 pills each time, 3 times a day, oral. Number of Cycles：4 weeks of treatment, the cured patients were followed up for 8 weeks to evaluate recurrence.
  Arms: Runzao zhiyang capsule
Drug: Runzaozhiyang capsule agent simulation — Runzaozhiyang capsule agent simulation：4 pills each time, 3 times a day, oral， Number of Cycles：4 weeks of treatment, the cured patients were followed up for 8 weeks to evaluate recurrence.
  Arms: Runzaozhiyang capsule agent simulation
Drug: Urea cream — Topical application, apply to the affected area and gently rub, 2 times a day.Number of Cycles：4 weeks of treatment, the cured patients were followed up for 8 weeks to evaluate recurrence.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Runzao zhiyang capsule in treating chronic eczema.

DETAILED DESCRIPTION:
Polygoni multiflori Preparata, dried rehmannia root, mulberry leaf, sophora flavescens, Honghuoma, for skin itching, acne, constipation due to blood vacuity and wind-dryness, also used in clinical treatment of eczema.

The purpose of this study is to evaluate the efficacy and safety of Runzao zhiyang capsule in treating chronic eczema.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with diagnostic criteria for chronic eczema(Referring to "the Chinese eczema diagnosis and treatment guidelines" in 2011);
* Investigator Global Assessment (IGA) score was 2 or 3;
* The skin lesions were localized, hypertrophy and dry, and the affected skin area was 3%~10% of body surface area (estimated by palm method); the diameter of target lesions was 2~10cm and located in the limbs or trunk.
* The course of chronic eczema is more than 6 months;
* Age 18 to 70, males or females;
* The Subjects obtain informed consent, participated the trial voluntarily. Procedure to obtain informed consent is in accordance with the provisions of Good Clinical Practise(GCP).

Exclusion Criteria:

* Subjects with acute eczema, subacute eczema, universal eczema, special type of eczema;
* Subjects used corticosteroids, immunosuppressive agents and ultraviolet irradiation in 4 weeks prior to the enrollment;
* Subjects were treated with antihistamine and topical drugs in 2 weeks;
* Women in Pregnancy, Lactation, or Planned pregnancy during the test;
* Comorbid with severe primary heart, liver, lung, kidney, blood disease, diabetes, thyroid disease or a serious disease affecting survival, such as cancer or HIV / AIDS;
* Subjects were allergic to test drug ingredients;
* Subjects could not give full informed consent because of mental and behavioral disorders;
* Suspected or identified with a history of alcohol or drug abuse;
* Have other diseases or conditions which may reduce the possibility of enrollment or complicate the recruiting process based on the investigator judgment. For example, working environment changed frequently led to easily lost follow-up;
* Have been or currently enrolled in other clinical trials within 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The efficiency(The number of cured cases and cases with marked effect) of disease： Using EASI score decline rate to judge. The decline rate of EASI = (before treatment EASI- After treatment EASI)/ before treatment EASI×100% | 0,4 weeks

SECONDARY OUTCOMES:
The decrease rate of EASI in each visit compare with baseline | 0,2,4,8,12 weeks
Changes in the degree of pruritus（test by visual analogue scale） in the follow-up visits compared with baseline | 0,2,4,8,12 weeks
DLQI (Dermatology Life Quality Index) score changes during the follow-up visits compared with baseline. | 0,2,4,8,12 weeks
The proportion of patients (EASI score greater than 10% of the patients before treatment) | 8,12 weeks
EASI score | 8,12 weeks

OTHER OUTCOMES:
Safety assessments will be based on adverse event reports. | 2,4,8,12 weeks
Safety assessments will be based on electrocardiogram, physical examinations, and clinical laboratory tests. | 0,2,4，8，12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gu heng, M.D., Principal Investigator — Dermotology hospital, Chinese academy of medical science
Locations (9):
- China (9):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqin Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-Sen Memorial Hospital,Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Dermotology hospital, Chinese academy of medical science, Nanjing, Jiangsu
  - Dermatology Hospital in Shandong Province, Jinan, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality